CLINICAL TRIAL: NCT05534633
Title: APPROACH 2.0: HIV, HCV and Syphilis Testing Through Pharmacies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Deborah Kelly, Professor, Memorial University of Newfoundland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HREB-2022.060
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections; HCV Infection; Syphilis Infection
MeSH Terms: conditions — HIV Infections; Hepatitis C

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants requesting test(s) for HIV, HCV, and/or syphilis (Other)
  Interventions: Other: Choice of STBBI test(s)

INTERVENTIONS:
Other: Choice of STBBI test(s) — Participants may receive a point of care HIV test, and/or point of care HCV test, and/or dry blood spot test, which can test for HIV, HCV, and syphilis, at the participants' choice.

SUMMARY:
Human Immunodeficiency Virus (HIV), hepatitis C (HCV), and syphilis are sexually transmitted and blood borne infections (STBBI) that affect millions of people worldwide and rates are rising in Canada. HCV and syphilis are curable, and HIV is treatable with virtually no risk of transmission to sexual partners when the infection is controlled, however, these outcomes require adequate testing. Unfortunately, an estimated 44% of Canadians living with HCV and 13% living with HIV are not diagnosed. These undiagnosed cases are the source of over half of new HIV infections. Furthermore, HIV-syphilis coinfection is common. Accessible testing forms a key pillar of an elimination strategy and acts as an access point for linking people to care. Community pharmacies are more accessible site for STBBI testing, compared to hospitals and doctors' offices. This is especially true for members of marginalized communities, some of whom are at higher risk of infection. The COVID-19 pandemic highlighted the need for low-barrier STBBI testing, as in-person healthcare services at doctors' offices and traditional screening clinics were scaled back. Pharmacies remained open throughout the pandemic.

The APPROACH 2.0 study will assess the impact of a pharmacy-based testing program for HIV, hepatitis C, and syphilis in participating pharmacies in three Canadian provinces: Newfoundland & Labrador, Alberta, and Nova Scotia on finding new diagnoses and linkages with care. Participants will be offered point of care tests for HIV and/or HCV and/or a dry blood spot test which will test for HIV, HCV, and syphilis. These tests are easy to administer. Results from the point of care tests are available immediately during the pharmacy visit while participants will be contacted with dried blood spot test results when available (approximately 2 weeks). Participants with reactive tests are linked with confirmatory testing and care, and those with non-reactive results are offered preventative services including HIV PrEP (as indicated) and counselling.

This study builds on a pilot study completed in 2017 (www.APPROACHstudy.ca).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older, speaks English, has provincial health card number, and is able and willing to provide informed consent.

Exclusion Criteria:

* Unwilling or unable to provide informed consent. Participants who have been previously diagnosed with HIV infection will not be eligible for HIV testing (point of care test or dry blood spot test). Participants who have previously been diagnosed with HCV are not eligible for HCV point of care test, but may request a dry blood spot test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of new HIV infections found through pharmacy testing in each province | Collected at the end of the study period (approximately one year)
Number and proportion of new HCV infections found through pharmacy testing in each province | Collected at the end of the study period (approximately one year)
Number and proportion of new syphilis infections found through pharmacy testing in each province | Collected at the end of the study period (approximately one year)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No